CLINICAL TRIAL: NCT06935214
Title: The Repeatability of the Effect of Caffeine Supplementation on Submaximal Physiological Responses and Cycling Time Trial Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SMU_ETHICS_2024-25_992
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Caffeine
Keywords: caffeine; genetics; cycling; time trial
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): 5 mg/kg dose of caffeine (in pill form) - Trial 1
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): 5 mg/kg dose of placebo (Maltodextrin in pill form) - Trial 2
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — 5 mg/kg of caffeine in pill form
  Arms: Caffeine
Dietary Supplement: Placebo — 5 mg/kg dose of maltodextrin in pill form
  Arms: Placebo
Dietary Supplement: Caffeine — 5 mg/kg dose of caffeine in pill form
  Arms: Caffeine

SUMMARY:
Recently, Grgic (2018) discussed the concept of responders and non-responders to caffeine supplementation highlighting the importance of the repeatability of results. However, the number of studies that have investigated this idea by repeating the same time-trial performance test multiple times with the same caffeine dose is sparse (Astorino et al., 2012; Del Coso et al., 2019). Furthermore, studies have shown that differences in the CYP1A2 genotype may account for some of the variation in time-trial performance (Guest et al., 2018). Thus, the current study aims to identify whether the effects of moderate caffeine supplementation (5 mg/kg) on time-trial performance are repeatable to aid the identification of responders and non-responders. Additionally, the study aims to determine if the CYP1A2 genotype may explain any of the variability in time-trial performance in trained male cyclists.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for inclusion in the study, participants must be regular cyclists, between 18 and 35 years of age, capable of completing a 20 km cycling time trial at a minimum speed of 30 km/h (arbitrary inclusion criteria to ensure a sufficient standard of athlete).

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood lactate concentration | From baseline to completion, up to 31 days
  Description: Change from baseline in blood lactate concentration measured at rest and at six different exercise intensities (55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate measured at rest and at seven different exercise intensities (55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer.
Oxygen uptake | From baseline to completion, up to 31 days
  Change from baseline in oxygen uptake measured at rest and at seven different exercise intensities (55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Perceived exertion | From baseline to completion, up to 31 days
  Change from baseline in rating of perceived exertion measured (using the 6-20 Borg scale) at seven different exercise intensities (55, 60, 65, 70, 75, and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer
Time trial completion time | From baseline to completion, up to 31 days
  Change from baseline in time to complete a time trial at a target amount of work on an electromagnetically-braked cycle ergometer calculated from the power output at maximal oxygen uptake and designed to last approximately 25 minutes.